CLINICAL TRIAL: NCT03824145
Title: Every Day Counts: A Lifestyle Program for Women With Metastatic Breast Cancer
Acronym: EDC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Loyola University Chicago (Other)
Responsible Party: Principal Investigator, Melinda Stolley, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 27600
Record Dates: First submitted 2018-02-19; First posted 2019-01-31 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Attention Control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention (Experimental): The experimental arm will receive a 16-week lifestyle intervention that promotes nutritional and physical activity changes concordant with those contained in the ACS nutrition and physical activity guidelines for cancer survivors. The 16-week intervention includes:
  1) a curriculum binder covering weekly topics and including self-monitoring tools to support adherence; 2) lifestyle coaching for 16-weeks, with in-person or virtual supervised exercise sessions and telephone-based sessions; 3) exercise supplies (Fitbit, resistance bands), 4) twice weekly text messaging targeting self-efficacy and social support; and 5) attendance to cooking classes emphasizing plant-based eating.
  Interventions: Behavioral: Lifestyle Intervention
- Attention Control (Other): The attention control participants will receive a home/work organization intervention:
  * Participants will receive a book with overview of home/work organization program with 16 weekly topics with an overview of each chapter.
  * Virtual or weekly phone calls- with a home organization coach with standard prompts.
  * Text messages supporting home/work organization.
  Following completion of the attention control home/work organization program and 16-week assessment, women will receive the lifestyle program.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The lifestyle intervention is a 16-week cognitive-behavioral intervention that addresses key changes in diet and PA behaviors to promote positive body composition changes.
  Arms: Immediate Intervention
Behavioral: Attention Control — The attention control participants will receive a home/work organization intervention:
  Following completion of the attention control home/work organization program and 16-week assessment, women will receive the lifestyle program.
  Arms: Attention Control

SUMMARY:
This multi-site study is being conducted to examine dietary and activity patterns, body composition, blood and quality of life in breast cancer patients. The study will recruit 176 women with MBC in Milwaukee (n=88) and Chicago (n=88).

DETAILED DESCRIPTION:
Aims/Objectives

Aim 1. To examine the efficacy of the Every Day Counts intervention in producing significant post-intervention changes in multidimensional QOL in women with MBC.

Hypothesis 1: Women randomized to the immediate EDC intervention (n=88) will exhibit greater improvements in multidimensional QOL compared to women randomized to the attention control (n=88).

Aim 2. To investigate the mechanistic effects of the Every Day Counts intervention on body composition, adipokines, serum biomarkers of inflammation and insulin sensitivity.

Hypothesis 2: The EDC intervention leads to improved QOL through mediating factors including body composition, prognostic serum biomarkers of inflammation and/or insulin resistance.

Exploratory Aim 3: To explore if microRNA (miRNA) signatures associated with inflammation and/or Metabolomics are altered with the EDC intervention.

Hypothesis: miRNAs identified in our pilot study (miR-10a-5p, miR-205-5p, and miR-211-5p) that regulate inflammation and/or Metabolomics will be related to QOL improvements and can identify women more likely to respond to lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years), female
* Confirmed Metastatic Breast Cancer
* Patients clinically stable with treated brain metastases are eligible
* Written documentation from their oncologist permitting study participation
* Determined to be "clinically stable" by their medical oncologist (i.e., no unintentional weight loss, no new symptoms or change in performance status for the past 4 weeks, no clinical [including laboratory] or radiologic evidence of disease progression, no recent or planned change in anti-neoplastic therapies, no reports of severe pain [≥ Grade 3 per the NCI CTCAE)
* Life expectancy >6 months

  -Written documentation from their oncologist permitting study participation
* Access to a mobile phone
* Understand/speak English fluently.
* Non-adherence to ACS nutritional or PA guidelines for cancer survivors as documented by questionnaire.

Exclusion Criteria:

* Does not meet the above criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Intervention adherence | 4 months
  Number of lifestyle coaching sessions completed out of a possible total of 16 sessions
Intervention retention | 4 months
  Number of women who complete the 4-month data collection
Intervention retention | 8 months
  Number of women who complete the 8-month data collection
Change in Quality of Life | Change from baseline to 4 months
  Patient reported outcomes as measured by Functional Assessment of Cancer Therapy-Measured by the Functional Assessment of Cancer Therapies Breast, Fatigue and Endocrine Symptoms (FACT-B, F and ES). The FACT-G is the overarching measure with a score range of 0-108; FACT-B (breast) subscale score range is 0-40; FACT-ES (endocrine symptoms) subscale score range is 0-76; FACT-F (fatigue) subscale is 0-52. Higher scores are better.
Change in Quality of Life | change from baseline to 8 months
  Patient reported outcomes as measured by Functional Assessment of Cancer Therapy-Measured by the Functional Assessment of Cancer Therapies Breast, Fatigue and Endocrine Symptoms (FACT-B, F and ES). The FACT-G is the overarching measure with a score range of 0-108; FACT-B (breast) subscale score range is 0-40; FACT-ES (endocrine symptoms) subscale score range is 0-76; FACT-F (fatigue) subscale is 0-52. Higher scores are better.
Body composition | change from baseline to 4 months
  Ratio of percent lean mass to percent adiposity as measured by DEXA. More lean mass and less adiposity is favorable.
Body composition | change from baseline to 8 months
  Ratio of percent lean mass to percent adiposity as measured by DEXA. More lean mass and less adiposity is favorable.

SECONDARY OUTCOMES:
Serum Biomarker Inflammation - C-Reactive Protein | Change from baseline to 4 month
  Analyzed by EVE technologies using standard ELISA kits
Serum Biomarker Insulin Resistance - Insulin | Change from baseline to 4 month
  Analyzed by EVE technologies using standard ELISA kits
Serum Biomarker Insulin Resistance- Glucose | Change from baseline to 4 month
  Analyzed by EVE technologies using standard ELISA kits
Serum Biomarker Inflammation - Tumor Necrosis Factor - alpha | Change from baseline to 4 month
  Analyzed by EVE technologies using standard ELISA kits
Serum Biomarker Insulin Resistance- C-Peptide | Change from baseline to 4 month
  Analyzed by EVE technologies using standard ELISA kits
Serum Biomarker Adipokine Dysregulation - Adiponectin | Change from baseline to 4 month
  Analyzed by EVE technologies using standard ELISA kits
Serum Biomarker Adipokine Dysregulation - Leptin | Change from baseline to 4 month
  Analyzed by EVE technologies using standard ELISA kits
Serum Biomarker Inflammation - Interleukin 6 | Change from baseline to 4 month
  Analyzed by EVE technologies using standard ELISA kits

OTHER OUTCOMES:
nRNA and Metabolomics - exploratory | Baseline to 3 months
  MTo explore if microRNA (miRNA) signatures associated with inflammation and/or Metabolomics are altered with the EDC intervention. analyzed using a Seahorse Bioscience extracellular flux analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Stolley, PhD, Principal Investigator — Principal Investigator
Locations (2):
- United States (2):
  - Loyola University, Maywood, Illinois
  - Medical College of Wisconsin, Milwaukee, Wisconsin